CLINICAL TRIAL: NCT05846984
Title: Learning Skills Together: A Randomized Controlled Trial of a Complex Care Skills Intervention to Improve AD/ADRD Caregiver Self-Efficacy
Brief Title: Learning Skills Together Family Caregiver Complex Intervention
Acronym: LST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kylie Meyer, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20220947; R01AG077554 (NIH)
Record Dates: First submitted 2023-04-01; First posted 2023-05-06 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Dementia; Alzheimer Disease; Caregiver Burden; Self Efficacy
MeSH Terms: conditions — Dementia; Alzheimer Disease; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In this study, participants, intervention facilitators, and the PI will be unblinded. Individuals collecting follow up surveys will be blinded to treatment condition, as will the study's statistician and data manager.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Learning Skills Together Intervention (Experimental): Complex care psychoeducation training intervention for family caregivers
  Interventions: Behavioral: Learning Skills Together Intervention
- Caregiver Healthy Living Intervention (Active Comparator): Healthy living intervention for family caregivers
  Interventions: Behavioral: Caregiver Healthy Living Intervention

INTERVENTIONS:
Behavioral: Learning Skills Together Intervention — Learning Skills Together is a 6-week psychoeducational intervention developed to improve caregivers' confidence when completing complex care tasks (e.g., using a gait belt). Participants are asked to attend six 1.5-hour Zoom-delivered group discussion sessions once per week, which cover topics such as how to communicate with someone who is living with dementia, medication management, and home safety. Participants are also provided with a workbook that accompanies each lesson, and includes short readings, videos, additional resources, as well as weekly practice and reflection exercises.
  Arms: Learning Skills Together Intervention
Behavioral: Caregiver Healthy Living Intervention — Participants in the Caregiver Healthy Living Intervention will participate in a 6-week educational intervention to help improve caregiver health behaviors (e.g., getting enough sleep). Participants are asked to attend six 1.5-hour Zoom-delivered group discussion sessions once per week, which cover topics such as how to eat a healthy diet, getting enough physical activity, and taking care of mental health. Participants are also provided a workbook that includes short readings and additional resources.
  Arms: Caregiver Healthy Living Intervention

SUMMARY:
Learning Skills Together (LST) is a 6-week psychoeducational intervention focused on complex care (nursing) tasks completed by family caregivers to persons living with Alzheimer's Disease and related dementias. This study aims to test the efficacy of LST at reducing caregiver depression and negative appraisal of behavioral symptoms of dementia by building caregiver self-efficacy. To do this, eligible participants will be randomized into an intervention group (LST) or a control group condition focused on healthy living for family caregivers. Participants will be asked to complete surveys before and after participating in the intervention or the control condition to determine whether change in hypothesized outcomes can be attributed to the intervention condition.

ELIGIBILITY:
Inclusion Criteria:

* Is aged 18 years or older
* Be a family member, including "families of choice," to an individual living with Alzheimer's disease or a related dementia who has received a diagnosis from a physician
* Provide assistance with at least two instrumental activities of daily living or one activity of daily living
* Report a Global Deterioration Scale (GDS) rating for care recipients between 4 to 6
* Commit to attending at least 5 of the 6 discussion sessions
* Has reliable access to the internet and email and be able to attend synchronous sessions using the Zoom videoconferencing platform

Exclusion Criteria:

* Unable to read and speak English
* Participated in Learning Skills Together in the past
* Plans to place the care recipient in a skilled nursing facility within the next 9 months (i.e., study duration)
* Was diagnosed with depression and/or started or significantly altered their depression treatment, including starting a pharmacological therapy or beginning therapy, in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Caregiver Self-Efficacy | Change from baseline to post-intervention survey 1 (within 2 weeks of completion); change from baseline to post-intervention survey 2 (3 months post-intervention); change from baseline to post-intervention survey 3 (6 months post-intervention)
  Self-efficacy will be measured using the 8-item Caregiver Self-Efficacy Scale (CSES-8; α=0.88 to 0.89; Ritter et al., 2020) Participants are asked to rate on a scale of 1 to 10 how confident they are with 8 aspects of caregiving (e.g., controlling upsetting thoughts). Scores range from 8 to 80, where higher scores indicate higher levels of caregiver self-efficacy. The outcome measure will use the average change score from baseline scores until each post-intervention survey (i.e., post-intervention, 3 months post-intervention, 6 months post-intervention).
Change in Caregiver Self-Efficacy with Complex Care (Author Generated) | Change from baseline to post-intervention survey 1 (within 2 weeks of completion); change from baseline to post-intervention survey 2 (3 months post-intervention); change from baseline to post-intervention survey 3 (6 months post-intervention)
  The investigators developed a caregiver complex care self-efficacy measure based upon discussions with healthcare faculty (Meyer et al., 2022). This 16-item scale asks about how confident caregivers feel with various complex care tasks (e.g., "Managing incontinence issues") and asks caregivers to rate their confidence from 0 ("Not at all confident") to 5 ("Very confident"). Pilot data showed high internal consistency (α=0.89). Higher scores indicate higher levels of self-efficacy with complex care tasks. The outcome measure will use the average change score from baseline scores until each post-intervention survey (i.e., post-intervention, 3 months post-intervention, 6 months post-intervention).
Change in Caregiver Self-Efficacy with Complex Care | Change from baseline to post-intervention survey 1 (within 2 weeks of completion); change from baseline to post-intervention survey 2 (3 months post-intervention); change from baseline to post-intervention survey 3 (6 months post-intervention)
  Self-efficacy with complex care will also be measured using the Caregiver Confidence in Sign/Symptom Management Scale (α=0.91), which subscales for Knowledge of Symptoms (α=0.56), Management of Cognitive Symptoms (α=0.82), Management of Medical Symptoms (α=0.78), and General Medical Management (α=0.94). Caregivers are asked how "true" statements are regarding their 1) knowledge, 2) ability to care for, and 3) make decisions about complex care tasks, as well as their level of confidence with various tasks. Scores range from 25 to 125, where higher scores indicate higher levels of caregiver self-efficacy with complex care. The outcome measure will use the average change score from baseline scores until each post-intervention survey (i.e., post-intervention, 3 months post-intervention, 6 months post-intervention).

SECONDARY OUTCOMES:
Change in Caregiver Resourcefulness | Change from baseline to post-intervention survey 1 (within 2 weeks of completion); change from baseline to post-intervention survey 2 (3 months post-intervention); change from baseline to post-intervention survey 3 (6 months post-intervention)
  Resourcefulness is measured using the 28-item Caregiver Resourcefulness Scale (α=0.85; Zauszniewski, 2006). This scale has two factors: one focused on help-seeking and another on self-help. Caregivers are asked the frequency at which they use different strategies to manage challenges, and may respond: Not at all like me (0), Pretty much not like me (1), A little bit not like me (2), A little bit like me (3), Pretty much like much like me (4), or Very much like me (5). Items are added together to create a total score. Scores range from 0 to 140, where higher scores indicate higher levels of resourcefulness. The outcome measure will use the average change score from baseline scores until each post-intervention survey (i.e., post-intervention, 3 months post-intervention, 6 months post-intervention).
Change in Caregiver Depressive Symptomology | Change from baseline to post-intervention survey 1 (within 2 weeks of completion); change from baseline to post-intervention survey 2 (3 months post-intervention); change from baseline to post-intervention survey 3 (6 months post-intervention)
  Depression will be measured with the Patient Health Questionnaire-9 (PHQ-9). (Kroenke et al., 2001) The PHQ-9 demonstrates specificity and sensitivity at 74-88% and 88-91%, respectively, for major depression with a cutoff score of 10. (Arroll et al., 2010; Kroenke et al., 2001). Scores range from 0 to 27, where higher scores indicate higher levels of depressive symptomology. The outcome measure will use the average change score from baseline scores until each post-intervention survey (i.e., post-intervention, 3 months post-intervention, 6 months post-intervention).
Appraisal of Behavioral Symptoms of Dementia | Change from baseline to post-intervention survey 1 (within 2 weeks of completion); change from baseline to post-intervention survey 2 (3 months post-intervention); change from baseline to post-intervention survey 3 (6 months post-intervention)
  Appraisal of behavioral symptoms of dementia will be measured with the Revised Memory and Behavior Checklist (RMBC). The RMBC includes 24-items and asks about caregiver appraisal of behavioral and psychological symptoms of dementia (e.g., Talking loudly or rapidly; α=0.90; Teri et al., 1992). Participants may indicate whether they feel Extremely bothered or upset, Very much bothered or upset, Moderately bothered or upset, A little bothered or upset, Not at all bothered or upset, Did not occur in the past week. Scores range from 0 to 96, wherein higher scores indicate higher levels of bother (more negative appraisal of behavioral symptoms of dementia). The outcome measure will use the average change score from baseline scores until each post-intervention survey (i.e., post-intervention, 3 months post-intervention, 6 months post-intervention).
Change in Quality of Care | Change from baseline to post-intervention survey 1 (within 2 weeks of completion); change from baseline to post-intervention survey 2 (3 months post-intervention); change from baseline to post-intervention survey 3 (6 months post-intervention)
  Quality of caregiving will be measured with the Task Management Strategy Index (TMSI; α=0.74 to 0.81; McClendon & Smyth, 2013). The 19-item TMSI was developed to assess caregivers' ability to manage their family member's functional disabilities. (Gitlin et al., 2002) Caregivers are asked how often they engage in strategies that support quality care. Caregivers indicate Never, Rarely, Sometimes, Often, or Always. Scores range from 19 to 95. Higher scores indicate higher quality of caregiving. The outcome measure will use the average change score from baseline scores until the post-intervention survey. The outcome measure will use the average change score from baseline scores until each post-intervention survey (i.e., post-intervention, 3 months post-intervention, 6 months post-intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Kylie N Meyer, PhD, Mac, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share de-identified research data collected from the Learning Skills Together clinical trial by depositing these data at the National Archive of Computerized Data on Aging (NACDA). De-identified data includes demographic information collected at baseline, survey data such as psychosocial outcome data, intervention participation/exposure, and other study-related data, including those published and unpublished by the investigator team. Documentation, such as code names and original survey questions, will also be uploaded to the repository in compliance with NACDA requirements (e.g., code names usable across software packages). We will also document meta-data (e.g., study title, investigator team). While uploading, we will note any transformations applied to the data, and will include both raw and transformed variables. Data will be shared in a .csv file, and documentation will be provided in PDF format.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified data will be deposited into NACDA repository as soon as possible but no later than within one year of the completion of the funded project period for the parent award or upon acceptance of the data for publication or public disclosure of a submitted patent application, whichever is earlier.
Access Criteria: Data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and could be used for secondary study purposes (e.g., cross-sectional analysis of baseline data). Novice users (e.g., doctoral students without advisor support) will have access to de-identified data and documentation regardless of level of experience or credentials. Sharing of analytic code will be provided at the discretion of the investigator team, based on the assessed qualification of the access requester, where "expert users" with an advanced academic degree or other relevant experience will be provided with code files.
URL: http://www.icpsr.umich.edu/web/pages/NACDA/index.html

REFERENCES:
- [Background] Arroll B, Goodyear-Smith F, Crengle S, Gunn J, Kerse N, Fishman T, Falloon K, Hatcher S. Validation of PHQ-2 and PHQ-9 to screen for major depression in the primary care population. Ann Fam Med. 2010 Jul-Aug;8(4):348-53. doi: 10.1370/afm.1139. PMID 20644190
- [Background] Gitlin LN, Winter L, Dennis MP, Corcoran M, Schinfeld S, Hauck WW. Strategies used by families to simplify tasks for individuals with Alzheimer's disease and related disorders: psychometric analysis of the Task Management Strategy Index (TMSI). Gerontologist. 2002 Feb;42(1):61-9. doi: 10.1093/geront/42.1.61. PMID 11815700
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] McClendon MJ, Smyth KA. Quality of informal care for persons with dementia: dimensions and correlates. Aging Ment Health. 2013;17(8):1003-15. doi: 10.1080/13607863.2013.805400. Epub 2013 Jun 11. PMID 24171485
- [Background] Meyer K, Glassner A, Norman R, James D, Sculley R, LealVasquez L, Hepburn K, Liu J, White C. Caregiver self-efficacy improves following complex care training: Results from the Learning Skills Together pilot study. Geriatr Nurs. 2022 May-Jun;45:147-152. doi: 10.1016/j.gerinurse.2022.03.013. Epub 2022 Apr 18. PMID 35447558
- [Background] Ritter PL, Sheth K, Stewart AL, Gallagher-Thompson D, Lorig K. Development and Evaluation of the Eight-Item Caregiver Self-Efficacy Scale (CSES-8). Gerontologist. 2022 Mar 28;62(3):e140-e149. doi: 10.1093/geront/gnaa174. PMID 33146727
- [Background] Teri L, Truax P, Logsdon R, Uomoto J, Zarit S, Vitaliano PP. Assessment of behavioral problems in dementia: the revised memory and behavior problems checklist. Psychol Aging. 1992 Dec;7(4):622-31. doi: 10.1037//0882-7974.7.4.622. PMID 1466831
- [Background] Zauszniewski JA. Resourcefulness. West J Nurs Res. 2016 Dec;38(12):1551-1553. doi: 10.1177/0193945916665079. No abstract available. PMID 27794127
- [Background] Zauszniewski JA, Burant CJ. Resourcefulness as a Mediator of the Effects of Dementia Symptoms and Caregiver Reactions on Caregiver Mental Health. Issues Ment Health Nurs. 2020 Jun;41(6):486-493. doi: 10.1080/01612840.2019.1693670. Epub 2020 Apr 7. PMID 32255406
- [Background] Zauszniewski JA, Lai CY, Tithiphontumrong S. Development and testing of the Resourcefulness Scale for Older Adults. J Nurs Meas. 2006 Spring-Summer;14(1):57-68. doi: 10.1891/jnum.14.1.57. PMID 16764178
- [Derived] Meyer K, Lee K, Thorngthip S, Burant P, Lippe M, Neidre D, White C, Norman R, Choi BY, Glover CM, Bell J, Hepburn K. A randomised controlled trial of the Learning Skills Together (LST) intervention to improve dementia family caregivers' self-efficacy with complex care. Trials. 2024 Jun 8;25(1):369. doi: 10.1186/s13063-024-08204-8. PMID 38851719